CLINICAL TRIAL: NCT00490659
Title: A Phase II Trial of Perioperative Chemotherapy (Gemcitabine and Cisplatin) and Adjuvant Chemoradiotherapy (-With Weekly Low-Dose Gemcitabine) in the Treatment of Nodes Positive NSCLC Patients
Brief Title: Trial of Perioperative Chemotherapy (Gemcitabine and Cisplatin) and Adjuvant Chemoradiotherapy (With Weekly Low Dose Gemcitabine) in Patients With Lung Cancer With Positive Nodes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8191; B9E-MC-S339
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: gemcitabine
Drug: cisplatin
Procedure: radical surgery
Procedure: chemoradiotherapy

SUMMARY:
The purpose of this study is to test feasibility, toxicity and efficacy of two different adjuvant treatment schedules in Stage II-IIIa Non-small cell lung cancer patients with positive lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC (any subtype). For patients entering Arm B is also allowed to confirm histopathological diagnosis of NSCLC intraoperatively during this trial.
* Node positive (clinically or pathologically) stage II disease or Stage IIIA: T1N1 or T2N1 or T1N2 or T2N2 or T3N1 or T3 N2, according to the revision by Mountain CF of American Joint Committee on Cancer (Mountain CF 1997, Fleming ID et al. 1997). For patient entering Arm B (with N0 stage) confirmation of N1-N2 stage must be obtained from intraoperative or post-surgery pathology report.
* Tumor amenable to curative surgical resection.
* Patients with clinically measurable lesions will be enrolled in this study. Measurability is determined according to RECIST criteria.

  • Pathological evaluation is performed after mediastinoscopy or after surgery
* No prior tumor therapy (surgery, radiotherapy, chemotherapy, immunotherapy, molecular targeted therapy, or any other type of tumor therapy).

Exclusion Criteria:

* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumor therapy, including radiotherapy, cytotoxic chemotherapy, immunotherapy, molecular target therapy.
* Serious concomitant disorders (for example, heart failure, poorly controlled diabetes) at the investigator's discretion.
* Presence of an uncontrolled, active infection requiring therapy (at the discretion of investigator.).
* Stage IIIb or IV.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-09; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
2-year overall survival

SECONDARY OUTCOMES:
Toxicity assessment
Assessment of feasibility of two treatment orders
Clinical and pathological response rate to neoadjuvant chemotherapy
Disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin, Poland

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com